CLINICAL TRIAL: NCT02205307
Title: A Randomized, Controlled, Parallel, Multicenter Study Assessing Perfusion Outcomes With PINPOINT® Near Infrared Fluorescence Imaging in Low Anterior Resection
Brief Title: A Study Assessing Perfusion Outcomes With PINPOINT® Near Infrared Fluorescence Imaging in Low Anterior Resection
Acronym: PILLAR III
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP PLR 03
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Rectal Cancer; Rectosigmoid Cancer
Keywords: Rectal cancer; Rectal neoplasm; Colorectal surgery; Anastomosis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PINPOINT or SPY Elite (Experimental): A low anterior resection will be performed according to the surgeon's standard practice with the addition of intraoperative imaging using PINPOINT near infrared fluorescence imaging or SPY Elite intraoperative imaging to assess colon and rectal tissue perfusion
  Interventions: Device: PINPOINT; Device: SPY Elite
- STANDARD (No Intervention): A low anterior resection will be performed according to the surgeon's standard practice

INTERVENTIONS:
Device: PINPOINT
  Arms: PINPOINT or SPY Elite
Device: SPY Elite
  Arms: PINPOINT or SPY Elite

SUMMARY:
This is a randomized, controlled, parallel, multicenter study to determine the difference in post-operative anastomotic leak rate in low anterior resection procedures where colon and rectal tissue perfusion is evaluated using PINPOINT as an adjunct to standard surgical practice compared to surgical procedures performed according to standard surgical practice alone.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Be undergoing open, or minimally invasive LAR for the treatment of a rectal or rectosigmoid neoplasm (Subjects with rectal or rectosigmoid neoplasm(s) may be treated with or without neoadjuvant therapy. Long-course neoadjuvant therapy must have been completed ≥6 weeks prior to LAR surgery (Day 0).
* Have a planned low circular stapled or transanally hand sewn anastomosis ≤10 cm from the anal verge.
* Have a colorectal or coloanal reconstruction with or without reservoir/pouch.
* Subjects who are women of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test at Day 0.
* Have signed an approved informed consent form for the study.
* Be willing to comply with the protocol.

Exclusion Criteria:

* Undergoing stapled anastomosis with the use of an experimental or non-FDA approved stapler.
* Undergoing ileoanal reconstruction, total colectomy or proctocolectomy, abdominoperineal resection, Hartmann's procedure, Hartmann's reversal or multiple synchronous colon resections (e.g., LAR and concomitant right colectomy).
* Has received and completed a course of pelvic radiotherapy ≥ 6 months prior to LAR surgery (Day 0).
* Has previously undergone a left sided colon resection.
* Has previously undergone a rectal resection.
* Has recurrent rectal or rectosigmoid cancer.
* Has a diagnosis of locally advanced rectal or rectosigmoid cancer undergoing extended en bloc operations.
* Has a diagnosis of Stage IV rectal or rectosigmoid cancer with any multifocal metastases or single site metastasis with tumor size of > 2 cm (Intraoperative incidental finding or preoperative suspicion of Stage IV cancer with isolated (single site) metastasis (≤ 2 cm) or limited metastases (≤3), with largest lesion ≤ 2 cm in size, does not exclude the subject).
* Has a diagnosis of inflammatory bowel disease (IBD). Subjects with rectal or rectosigmoid cancer neoplasms and IBD are excluded.
* Has hepatic dysfunction defined as Model for End-Stage Liver Disease (MELD) Score >12.
* Renal dysfunction defined as creatinine ≥ 2.0 mg/dL.
* Has known allergy or history of adverse reaction to ICG, iodine or iodine dyes.
* Has, in the Investigator's opinion, any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results.
* Is actively participating in another investigational clinical study which, in the Investigator's or Sponsor's opinion, would interfere in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2015-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Stamos, MD, Principal Investigator — University of California, Irvine; Steven Wexner, MD, Principal Investigator — Cleveland Clinic Florida
Locations (24):
- United States (24):
  - John Muir Medical Center, Concord Campus, Concord, California
  - Kaiser Permanente, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California, San Francisco, San Francisco, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barnes Jewish Medical Center, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Jafari MD, Pigazzi A, McLemore EC, Mutch MG, Haas E, Rasheid SH, Wait AD, Paquette IM, Bardakcioglu O, Safar B, Landmann RG, Varma MG, Maron DJ, Martz J, Bauer JJ, George VV, Fleshman JW Jr, Steele SR, Stamos MJ. Perfusion Assessment in Left-Sided/Low Anterior Resection (PILLAR III): A Randomized, Controlled, Parallel, Multicenter Study Assessing Perfusion Outcomes With PINPOINT Near-Infrared Fluorescence Imaging in Low Anterior Resection. Dis Colon Rectum. 2021 Aug 1;64(8):995-1002. doi: 10.1097/DCR.0000000000002007. PMID 33872284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PINPOINT or SPY Elite | STANDARD
Started | 178 | 169
Completed | 161 | 163
Not Completed | 17 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PINPOINT or SPY Elite | STANDARD | Total
Number analyzed (Participants) | 178 | 169 | 347
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean | 57.2 (11.14) | 56.5 (11.59) | 56.9 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 70 | 139
  Male | 109 | 99 | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 7 | 14 | 21
  Race/Ethnicity: African American | 23 | 14 | 37
  Race/Ethnicity: Hispanic | 23 | 14 | 37
  Race/Ethnicity: White | 123 | 122 | 245
  Race/Ethnicity: Other | 2 | 5 | 7
Height [Mean (Standard Deviation); unit: cm] | 171.89 (9.814) | 171.32 (9.790) | 171.61 (9.792)
Weight [Mean (Standard Deviation); unit: kg] | 82.49 (19.743) | 83.11 (19.815) | 82.79 (19.752)
Smoking Status [Count of Participants; unit: Participants]
  Yes | 52 | 31 | 83
  No | 126 | 138 | 264
Alcohol Consumption [Count of Participants; unit: Participants]
  Yes | 81 | 80 | 161
  No | 97 | 89 | 186
MELD Score (Model for End-Stage Liver Disease) [Mean (Standard Deviation); unit: units on a scale (6-40)] — The Model for End-Stage Liver Disease (MELD) consists of serum bilirubin, creatinine levels, International Normalized Ratio (INR) for prothrombin time, and Serum Sodium levels. Subjects with hepatic dysfunction defined as Model for End-Stage Liver Disease (MELD) Score >12 were excluded from the study. The MELD score can range from 6 to 40 with higher numbers indicating more severe disease.
  units on a scale (6-40) | 6.8 (1.06) | 6.7 (1.36) | 6.8 (1.22)
Long-Course Neoadjuvant Therapy [Count of Participants; unit: Participants]
  Yes | 113 | 111 | 224
  No | 65 | 58 | 123
Pre-Operative Diagnosis [Count of Participants; unit: Participants]
  Rectal Cancer | 144 | 143 | 287
  Rectosigmoid Cancer | 27 | 24 | 51
  Polyp | 3 | 1 | 4
  Other | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Anastomotic Leak Rate
Description: Anastomotic leak rate in low anterior resection procedures where colon and rectal tissue perfusion is evaluated using PINPOINT Endoscopic Fluorescence imaging or SPY Elite imaging as an adjunct to standard surgical practice compared to surgical procedures performed according to standard surgical practice alone.
Time Frame: Day 0 to Week 8 (+/- 2 weeks)
Population: Modified Intent-to-Treat (mITT): the mITT analysis population includes all randomized subjects in whom a low anterior resection surgical procedure is initiated or at least one injection with ICG was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | PINPOINT or SPY Elite | STANDARD
Number analyzed (Participants) | 175 | 168
Participants
  Subjects with Post-Operative Anastomotic Leak | 14 | 16
  Subjects Known to be Anastomotic Leak Free | 148 | 148
  Unknown/Lost to Follow Up | 13 | 4

2. Secondary Outcome: Rate of SPY Visualization and Tissue Perfusion
Description: The ability of PINPOINT or SPY Elite to provide sufficient visualization for assessment of blood flow and related tissue perfusion during the procedure
Time Frame: Day 0 (Day of Surgery)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PINPOINT or SPY Elite
Number analyzed (Participants) | 175
Participants | 167

3. Secondary Outcome: Incidence of Post-Operative Abscess Requiring Surgical Management
Description: Rate of postoperative abscess requiring surgical management.
Time Frame: Day 0 to Week 8 (+/- 2 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PINPOINT or SPY Elite | STANDARD
Number analyzed (Participants) | 175 | 168
Participants
  Yes | 10 | 7
  No | 165 | 161

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse events were monitored/assessed for all randomized subjects. 8 subjects were withdrawn after randomized and not treated either by SPY or STANDARD treatments.
Groups:
- Not Treated: Not treated by either perfusion (PINPOINT/SPY Elite) or standard treatment.
Arm/Group | PINPOINT or SPY Elite | STANDARD | Not Treated
All-Cause Mortality (participants affected / at risk) | 3/171 | 1/168 | 0/8
Serious Adverse Events (participants affected / at risk) | 44/171 | 52/168 | 0/8
Other Adverse Events (participants affected / at risk) | 155/171 | 146/168 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PINPOINT or SPY Elite (N=171) | STANDARD (N=168) | Not Treated (N=8)
Ileus (Gastrointestinal disorders) | 4 | 8 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 2 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Functional Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Internal Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intra-Abdominal Hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Anastomotic Leak (Injury, poisoning and procedural complications) | 7 | 8 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 2 | 2 | 0
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 2 | 0
Anastomotic Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision Site Erosion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ureteric Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic Abscess (Infections and infestations) | 2 | 4 | 0
Sepsis (Infections and infestations) | 2 | 2 | 0
Abdominal Abscess (Infections and infestations) | 0 | 3 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 8 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 2 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Arterial Haemorrhage (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 — Adverse Device Effect - classified as mild, suspected to be related to PINPOINT/ICG but not to the surgical procedure itself, was assessed as Grade II and resolved.
Ischaemia (Vascular disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Pelvic Haematoma (Reproductive system and breast disorders) | 2 | 0 | 0
Pelvic Fluid Collection (Reproductive system and breast disorders) | 1 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Death (General disorders) | 3 | 1 | 0
Multi-organ Failure (General disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Ileostomy Closure (Surgical and medical procedures) | 0 | 1 | 0
Small Intestinal Resection (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PINPOINT or SPY Elite (N=171) | STANDARD (N=168) | Not Treated (N=8)
Procedural Pain (Injury, poisoning and procedural complications) | 62 | 62 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 9 | 12 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 7 | 11 | 0
Nausea (Gastrointestinal disorders) | 45 | 41 | 0
Vomiting (Gastrointestinal disorders) | 22 | 29 | 1
Abdominal Pain (Gastrointestinal disorders) | 27 | 15 | 0
Abdominal Distension (Gastrointestinal disorders) | 12 | 16 | 0
Ileus (Gastrointestinal disorders) | 6 | 13 | 0
Pain (General disorders) | 21 | 11 | 0

LIMITATIONS AND CAVEATS:
The interpretation of the efficacy results is limited due to the fact that the study was stopped early, which may have adversely affected the statistical power of some tests.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT02205307/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT02205307/SAP_001.pdf